CLINICAL TRIAL: NCT00010179
Title: Randomized Phase II Study Of NX 211 Given By Two Different Intravenous Schedules In Advanced And/Or Recurrent Epithelial Ovarian Cancer
Brief Title: Lurtotecan Liposome in Treating Patients With Advanced or Recurrent Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I138; CAN-NCIC-IND138 (Other: PDQ); CDR0000068453 (Other: PDQ)
Record Dates: First submitted 2001-02-02; First posted 2004-02-26 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: lurtotecan liposome

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing of die.

PURPOSE: Randomized phase II trial to compare the effectiveness of two treatment regimens of lurtotecan liposome in patients who have advanced or recurrent ovarian epithelial cancer, primary fallopian tube cancer, or peritoneal cancer that has been previously treated with chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the anti-tumor efficacy of two treatment schedules of lurtotecan liposome, in terms of clinical/radiological response and CA125 tumor marker, in patients with previously treated advanced or recurrent ovarian epithelial cancer. II. Compare the safety, pharmacokinetics, and possible pharmacokinetic/pharmacodynamic relationships of these treatment schedules in these patients. III. Compare the time to progression in patients treated with these treatment schedules.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to time from last prior chemotherapy (less than 6 months vs 6 months or more) and number of prior chemotherapy regimens (1 vs 2). Patients are randomized to one of two treatment arms. Arm I: Patients receive lurtotecan liposome IV over 30 minutes on days 1-3. Arm II: Patients receive lurtotecan liposome IV over 30 minutes on days 1 and 8. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses after documented CR. Patients achieving partial response (PR) receive 4 additional courses after documented PR or until disease progression at investigator's discretion. Patients with stable disease continue therapy for a maximum of 6 courses. Patients are followed at 4 weeks and then every 3 months until disease relapse or progression.

PROJECTED ACCRUAL: A total of 40-74 patients (20-37 per treatment arm) will be accrued for this study within 10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed ovarian epithelial cancer Primary fallopian or peritoneal cancer allowed Clinically and/or radiologically documented advanced and/or recurrent disease At least one site of disease unidimensionally measurable: Minimum indicator lesion site as follows: At least 10 mm on spiral CT scan At least 20 mm on conventional CT scan At least 20 mm on chest x-ray or physical exam No recent prior radiotherapy to indicator lesion(s) Clear disease progression or new lesion within a previously irradiated field allowed Previously treated with one or two chemotherapy regimens At least one regimen must have contained cisplatin or carboplatin (changing from one prior platinum compound to another for disease progression or failure to respond is considered a second regimen) Use of same prior chemotherapy combination for first-line and second-line therapy is considered two regimens No borderline ovarian tumor No ascites as only disease presentation No abdominal adenocarcinoma of unknown origin No symptomatic brain metastasis that are potentially life-threatening or require active treatment

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST/ALT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No other prior malignancy within the past 5 years unless definitively treated with no evidence of recurrence No known hypersensitivity to systemic liposomal formulations or drugs chemically related to study drug No other serious illness or medical condition that would preclude study No active uncontrolled infection No complete bowel obstruction No history of significant neurologic or psychiatric disorder that would preclude informed consent Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosourea) and recovered No prior topotecan or other topoisomerase-I inhibitor No other concurrent cytotoxic therapy for ovarian cancer Endocrine therapy: No concurrent hormonal therapy for ovarian cancer Radiotherapy: See Disease Characteristics Recovered from prior radiotherapy At least 4 weeks since prior radiotherapy to area comprising at least 25% of bone marrow stores Surgery: At least 4 weeks since prior major surgery and recovered Other: At least 30 days since prior investigational agent or new anticancer therapy No other concurrent investigational therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2000-10-31 (Actual); Primary Completion 2002-10-22 (Actual); Study Completion 2008-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert N. Grimshaw, MD, Study Chair — Nova Scotia Cancer Centre
Locations (14):
- Canada (8):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - BCCC - Cancer Center for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Queen's University, Kingston, Ontario
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- United Kingdom (6):
  - City Hospital NHS Trust, Birmingham, England
  - Royal Marsden NHS Trust, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Weston Park Hospital, Sheffield, England
  - Beatson Oncology Centre, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dark GG, Calvert AH, Grimshaw R, Poole C, Swenerton K, Kaye S, Coleman R, Jayson G, Le T, Ellard S, Trudeau M, Vasey P, Hamilton M, Cameron T, Barrett E, Walsh W, McIntosh L, Eisenhauer EA. Randomized trial of two intravenous schedules of the topoisomerase I inhibitor liposomal lurtotecan in women with relapsed epithelial ovarian cancer: a trial of the national cancer institute of Canada clinical trials group. J Clin Oncol. 2005 Mar 20;23(9):1859-66. doi: 10.1200/JCO.2005.02.028. Epub 2005 Feb 7. PMID 15699482
- [Result] Calvert AH, Grimshaw R, Poole C, et al.: Randomized phase II trial of two intravenous schedules of the liposomal topoisomerase I inhibitor, NX211, in women with relapsed epithelial ovarian cancer (OVCA): an NCIC CTG study. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-830, 2002.
- [Result] Wolf J, Hamilton M, Eisenhauer E, et al.: Pharmacokinetics of NX211 (liposomal lurtotecan) using a limited sampling model in a phase II trial of patients with ovarian cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-485, 2002.